CLINICAL TRIAL: NCT00850733
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study of Safety and Efficacy of a Single Treatment With 2 Dose Levels of BOTOX Purified Neurotoxin Complex Followed by a Treatment With BOTOX in Patients With…
Brief Title: 516-BOTOX Urinary Incontinence Detrusor
Status: Completed | Type: Observational
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: Allergan (Industry)
Responsible Party: Michael Albo, MD, Veterans Medical Research Foundation
Other Study IDs: 071304; VMRF Project #07366
Record Dates: First submitted 2009-02-20; First posted 2009-02-25 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Urinary Incontinence; Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The specific aim of this study is to evaluate the safety and efficacy of each of 2 dosages of BOTOX® (200 U or 300 U) compared to placebo injected into the detrusor for the treatment of urinary incontinence caused by neurogenic detrusor overactivity in patients who have not been adequately managed with anticholinergic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female, aged 18 to 80 years old.
2. Patient weighs ≥ 50 kg (110 lb).
3. Patient has urinary incontinence as a result of neurogenic detrusor overactivity for a period of at least 3 months prior to screening as a result of spinal cord injury or multiple sclerosis, determined by documented patient history. In addition:

   * Spinal cord injury patients must have a stable neurological injury level at T1 or below (cervical injuries are excluded) occurring ≥ 6 months prior to screening.
   * Multiple sclerosis patients must be clinically stable in the investigator's opinion for ≥ 3 months prior to screening and have an Expanded Disability Status Scale score ≤ 6.5.
4. Patient has detrusor overactivity (defined as a phasic rise in bladder pressure during the filling phase determined by urodynamics) demonstrated during the screening period or Day 1 (prior to randomization).
5. Patient is able to complete study requirements including bladder diary completion and attend all study visits (telephone and clinic), in the opinion of the investigator.
6. Patient has not been adequately managed with one or more anticholinergics for their urinary incontinence, in the opinion of the investigator. Not adequately managed is defined as an inadequate response or intolerable side effects after at least one month of anticholinergic therapy on an optimized dose.
7. For patients taking anticholinergic medication for their neurogenic overactive bladder, dose is stable and patient is willing to maintain same dosing during study participation.
8. Patient has a negative pregnancy result if female and of childbearing potential.

   The following criteria are also required for entry into the study at Randomization/Day 1:
9. Patient experiences ≥ 14 episodes of urinary incontinence per week with no more than 2 incontinent-free days determined by completion of patient bladder diary during the screening period.
10. Patient currently uses or is willing to use clean intermittent catheterization (CIC) to empty the bladder (indwelling catheter is not permitted). Patients currently on CIC should be willing to maintain an established CIC frequency throughout the study. Caregiver may perform CIC.
11. Patients with a negative urine culture result must take an antibiotic medication for 3 days immediately prior to Randomization/Day 1 and agree to continue antibiotic medication for at least 3 days following treatment. Patients with a positive urine culture result indicating urinary tract infection (UTI) must take an antibiotic to which the identified organism is sensitive for at least 5 days immediately prior to Randomization/Day 1 and continue for 3 days following the procedure (or longer as needed) and patient is asymptomatic for UTI on day of treatment. A UTI is defined as either a positive urine culture result with a bacteriuria count of > 105 CFU/mL conjoint with a leukocyturia > 5/hpf at screening or a positive urine culture that, in the investigator's opinion, requires antibiotic therapy.

Exclusion Criteria:

1. Patient has history or evidence of any pelvic or urological abnormalities including but not limited to the following:

   * elevated serum creatinine > 2 times the upper limit of normal (reference range)
   * history of or current hematuria, 1) if the hematuria is determined to be a pathologic condition or 2) is uninvestigated
   * interstitial cystitis in the opinion of the investigator
   * bladder stones within 6 months of screening
   * surgery or bladder disease other than detrusor overactivity that may impact bladder function with the exception of surgeries for bladder stones (> 6 months) and stress incontinence, uterine prolapse, rectocele, or cystocele (>1 year) from screening
2. Patient has had previous or current botulinum toxin therapy of any serotype for any urological condition or, treatment within 3 months of Randomization/Day 1 for any other condition or use.
3. Patient has been immunized for any botulinum toxin serotype.
4. Patient discontinued anticholinergic medication for overactive bladder < 21 days prior to Randomization/Day 1.
5. Patient has a history or current diagnosis of bladder cancer or has urine cytology results which may indicate bladder cancer not ruled out by investigator at Randomization/Day 1. Suspicious urine cytology abnormalities require the investigator's assessment to ensure that the findings are not indicative of malignancy.
6. Patient is male with previous or current diagnosis of prostate cancer. Patients with a PSA level greater than 4.0 ng/mL will require a biopsy to rule out prostate cancer, unless a prostatic biopsy has been performed on the patient within the past 12 months.
7. Patient has 24 hour total volume voided > 3000 mL of urine determined by completion of patient bladder diary collected over one consecutive 24 hour period during the 7 day diary collection period prior to Randomization/Day1.
8. Patient has a post void residual volume above 200 mL for patients who micturate or have a mixed catheterization/spontaneous micturition pattern.
9. Patient has an active genital infection, other than genital warts, either concurrently or within 4 weeks prior to screening.
10. Patient uses any anti-platelet or anticoagulant therapy or is using medications with anti-coagulative effects within 3 days prior to treatment. Some medications may need to be withheld for > 3 days per clinical judgment of the investigator (refer to Section 8.2.2 Prohibited Medications/Treatments for details).
11. Patient has hemophilia or other clotting factor deficiencies or disorders that cause bleeding diatheses.
12. Patient has had concurrent treatment or treatment within 6 months of Randomization/Day 1 with capsaicin or resiniferatoxin.
13. Patient is currently using or plans to use an implanted or non-implantable electrostimulation/neuromodulation device for treatment of overactive bladder.
14. Patient has a known allergy or sensitivity to any components of the study medication, anesthetics or antibiotics or any other products associated with the treatment and general study procedures.
15. Patient has any medical condition that may put the patient at increased risk with exposure to BOTOX® including diagnosed myasthenia gravis, Eaton-Lambert syndrome or amyotrophic lateral sclerosis.
16. Patient is female and pregnant, nursing or planning a pregnancy during the study, or of childbearing potential and unable or unwilling to use a reliable form of contraception during the study.
17. Patient is currently or has previously participated in another therapeutic or device study within 30 days of screening.
18. Patient has any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit 260 patients nationwide with an expected recruitment of 6 patients at the VA San Diego Healthcare System. Patients must be between 18-80 years of age and will include patients with neurogenic detrusor overactivity as a result of spinal cord injury or multiple sclerosis, with urinary incontinence, who have not been adequately managed with anticholinergic therapy. 50% of the patients randomized will be of spinal cord injury etiology and 50% of multiple sclerosis etiology.
Sampling Method: Non-Probability Sample
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)